CLINICAL TRIAL: NCT02828683
Title: Safety and Efficacy of TCD-10023 (Ultimaster) Drug-eluting Stent in Management of Patients With Acute ST-Elevation Myocardial InfaRction - MASTER Study
Brief Title: Safety and Efficacy of TCD-10023 (Ultimaster) Drug-eluting Stent in STEMI Patients - MASTER Study
Acronym: MASTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T120E4
Record Dates: First submitted 2013-05-16; First posted 2016-07-12 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Acute ST Segment Elevation Myocardial Infarction
Keywords: DES; PCI; STEMI; Interventional Cardiology
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ultimaster, Drug Eluting Stent (Experimental): Primary PCI in patients with ST segment elevation myocardial infarction with a new Drug Eluting Stent, Ultimaster
  Interventions: Device: PCI in patients with ST-elevation myocardial infarction
- Kaname, Bare metal stent (Active Comparator): Primary PCI in patients with ST segment elevation myocardial infarction with a Bare Metal Stent - Kaname
  Interventions: Device: PCI in patients with ST-elevation myocardial infarction

INTERVENTIONS:
Device: PCI in patients with ST-elevation myocardial infarction — Percutaneous coronary intervention in patients with ST segment elevation myocardial infarction (STEMI)
  Other Names: Primary PCI
  Arms: Ultimaster, Drug Eluting Stent
Device: PCI in patients with ST-elevation myocardial infarction — Percutaneous coronary intervention in patients with ST-segment elevatio myocardial infarction
  Other Names: Primary PCI
  Arms: Kaname, Bare metal stent

SUMMARY:
The aim of the study is to demonstrate the safety and efficacy of the TCD-10023 (Ultimaster) sirolimus eluting stent in patients with acute ST-elevation myocardial infarction (STEMI), by proving superiority with respect to in-stent late loss at 6 months to the Kaname bare metal stent and non-inferiority with respect to Target Vessel Failure (TVF) at 12 months.

DETAILED DESCRIPTION:
MASTER is prospective, randomized (3:1), single blind, controlled, superiority (efficacy) and non-inferiority (safety and efficacy), multi center, two-arm trial of TCD-10023 (Ultimaster) drug eluting stent (test) and Kaname bare metal stent (comparator).

Patients will be followed at 30 days, 6, and 12 months post-procedure and annually for 3 years.

500 patients with clinical follow up will be randomized in 3:1 ratio (375 in TCD-10023 arm and 125 in Kaname arm). Among them, 100 patients will be randomized in the same, 3:1 ratio, to angiographic follow up at 6 months in preselected hospitals (75 in TCD-10023 and 25 in Kaname arm)

ELIGIBILITY:
Inclusion Criteria:

* Age equal or more than 18 years
* Chest pain > 20 minutes
* Primary PCI <24h from symptoms onset
* ST-segment elevation of > 1 mm in > 2 contiguous leads, or (presumably new) left bundle branch block, or true posterior MI with ST depression of > 1 mm in > 2 contiguous anterior leads
* Presence of at least one acute infarct artery target vessel with one or more coronary artery stenoses in a native coronary artery from 2.5-4.0 mm in diameter that can be covered with one or multiple stents
* Signed informed consent

Exclusion Criteria:

* Female of childbearing potential (age < 50 and last menstruation within the last 12 months), who did not underwent tubal ligation, ovariectomy or hysterectomy
* Known intolerance to aspirin, clopidogrel, heparin, bivalirudin, cobalt, chromium, nickel, sirolimus or contrast material
* Currently participating in another trial before reaching primary endpoint
* Mechanical complication of acute myocardial infarction (e.g. cardiogenic shock…)
* Acute myocardial infarction secondary to stent thrombosis
* Previously stented infarction related artery (IRA)
* Planned surgery within 6 months of PCI unless dual antiplatelet therapy is maintained throughout the peri-surgical period
* Patients with non-cardiac comorbid conditions with life expectancy< 1 year or that may result in protocol non-compliance
* History of bleeding diathesis or known coagulopathy
* Use of oral anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-07 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Target Vessel Failure (TVF) | 12 months
  Composite endpoint of cardiac death, target vessel myocardial infarctio and target vessel revascularization

SECONDARY OUTCOMES:
Target lesion failure | 1 month, 6 months, 12 months, 2 and 3 years
  Composite of cardiac death, target vessel myocardial infarction, target lesion revascularization 2. Target vessel failure (TVF) Comosite of cardiac death, target vessel myocardial infarction, target lesion revascularization
Target vessel failure | 1 month, 6 months, 2 and 3 years
  Composite of cardiac death, target vessel myocardial infarction, target vessel revascularization
Stent thrombosis | 1 month, 6 months, 12 months, 2 and 3 years
  Thrombosis in study stents
Patient oriented endpoint Composite of any death, any myocardial infarction, any coronary revascularization | 1 month, 6 months, 12 months, 2 and 3 years
  Composite of any death, any myocardial infarction, any coronary revascularization
Target lesion revascularization | 1 month, 6 months, 12 months, 2 and 3 years
  revascularization of treated lesion
Bleeding | 1 month, 6 months, 12 months, 2 and 3 years
  Access or non access site bleeding
Safety - revascularization, stroke, definite stent thrombosis or major bleeding | 1 month
  revascularization, stroke, definite stent thrombosis or major bleeding at 1 month
In-Stent late loss | 6-mnths
  angiographic assessment of late loss at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Borovicanin, MD, Study Director — Terumo Europe
Locations (13):
- Instituto Dante Pazzanese, São Paulo, Brazil
- Italy (4):
  - Azienda Ospedaliero Universitaria, Policlinico "Vittorio Emanuele" - Ospedale Ferrarotto, Catania
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Cardiologico Monzino, Milan
  - San Raffaele Hospital, Milan
- PHE University Cardiology clinic, Skopje, North Macedonia
- Serbia (3):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Zemun (CHC Zemun), Belgrade
  - Clinical center Nis (CCNIs), Niš
- Spain (4):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Virgen Arrixaca-Murcia, El Palmar
  - Hospital Universitario Central Asturias-Oviedo, Oviedo
  - Complejo Hospitalario Universitario Santiago de Compostela, Santiago de Compostela